CLINICAL TRIAL: NCT06233279
Title: Single-center, Double-blind, Placebo-controlled, Randomized Clinical Trials for Safety and Efficacy Assessment of Symptoms Related to Autism Spectrum Disorder Using NuEyne P01 in Patients With Autism Spectrum Disorder
Brief Title: Study of Application of Transcutaneous Trigeminal Nerve Stimulation on Autism Spectrum Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nu Eyne Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NE_PSY_001
Record Dates: First submitted 2023-11-08; First posted 2024-01-31 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2023-11

CONDITIONS: Autism Spectrum Disorder
Keywords: ASD
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Charge-Balanced, Symmetric Nerve Stimulation device is used during night sleep for eight hours each day for 4 weeks (28 days).
  Interventions: Device: Charge-Balanced, Symmetric Nerve Stimulation
- Control Group (Sham Comparator): Sham Stimulation device is used during night sleep for eight hours each day for 4 weeks (28 days).
  Interventions: Device: Sham Stimulation

INTERVENTIONS:
Device: Charge-Balanced, Symmetric Nerve Stimulation — Charge-Balanced, Symmetric Nerve Stimulation device is used during night sleep for eight hours each day for 4 weeks (28 days).
  Arms: Experimental Group
Device: Sham Stimulation — Sham Stimulation device is used during night sleep for eight hours each day for 4 weeks (28 days).
  Arms: Control Group

SUMMARY:
This study aims to evaluate the safety and the efficacy of applying transcutaneous trigeminal nerve stimulator (NuEyne P01) on autism spectrum disorder.

DETAILED DESCRIPTION:
Duration of study period (per participant): Screening period (-28~0 days), Intervention period (28 days) Patient needs to visit site at least 4 times (V1, V2, V4, V6). V2 can be done with V1. Tele-visit should be done on V3 (day 7), V5 (day 21).

ELIGIBILITY:
Inclusion Criteria:

* Children over 7 years old and under 12 years old
* Patients diagnosed with autism spectrum disorder
* A person who has a total intelligence index of 70 or higher and has no problems with basic language communication
* A person who agrees not to use any medical device other than this clinical trial medical device during the clinical trial period
* A person who does not take a concurrent drug from screening to the end of the study, or who can maintain the concurrent drug during the clinical trial period without any change or addition
* Voluntary written consent to participate in this clinical trial

Exclusion Criteria:

* Those who participated in other clinical trials within 30 days from the screening date
* If it is difficult to understand the contents of treatment due to the limitation of intelligence index or language ability, and if it is difficult to conduct a study
* When there is a risk of clinically significant behavioral problems, emotional control problems, psychiatric symptoms, self-harm, or other harm that can affect the treatment process
* Psychiatric hospitalization history
* A person with acute or chronic medical or mental illness
* A person with a history of seizures
* Serious trauma and surgery within 1 month
* A person who is deemed to have a problem with the adhesion of electrodes due to inflammatory reactions or other dermatological problems on the skin around the forehead to which electrodes of clinical trial medical devices are attached
* If it is need to take sleep medications [benzodiazepine, melatonin, trazodone] (*However, it is participated after having a washout period of at least two weeks.)
* A person who is deemed to have other reasons for prohibition of use of clinical trial medical devices (including heart-related problems, seizures, metal or electronic devices implanted in the head, people with unknown pain, pacemaker transplant, etc.)
* When it is determined by the researcher that it is difficult for the subject to continue voluntary participation in the study due to the lack of cooperation and motivation for treatment
* Other cases where it is deemed difficult to participate in the study by the researcher's judgment

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2022-11-15 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Safety evaluation | baseline, 4 weeks
  Occurrence of adverse events caused by the investigational device, including psychiatric abnormality, skin abnormality at the contact site, headache, sleepiness, trigeminal nerve abnormality, etc. is checked.

SECONDARY OUTCOMES:
Changes in Level of functioning | baseline, 4 weeks
  This is measured by two questionnaires, WISC-IV and Vineland Adaptation Behavior Scale-II, to confirm cognitive function. It is can be judged by combining the results of each questionnaire test.
  This clinical trial, as an exploratory clinical trial, aims at seeing whether there is a statistical difference between before and after the treatment in observation items. If both items are significant, cognitive function is considered significant.
Changes in Social reciprocity | [Time Frame: baseline, 2 weeks, 4 weeks]
  This is measured in five questionnaires, Aberrant Behavior Checklist-II (ABC-2), Autistic Quotient (AQ), Social Responsiveness Scale-2 (SRS-2), Korean Childhood autism rating scale (K-CARS-2), Social communication questionnaire (SCQ) to confirm sociality. It can be judged by combining the results of each questionnaire test. This clinical trial, as an exploratory clinical trial, aims at seeing whether there is a statistical difference between before and after the treatment in observation items.
  This clinical trial, as an exploratory clinical trial, aims at seeing whether there is a statistical difference between before and after the treatment in observation items. If more than three are significant, the Social reciprocity is considered significant. This result is judged to be significant as the result value is lower.
Changes in Executive function | baseline, 2 weeks, 4 weeks
  This is measured in five questionnaires, Children's color trail making test 1 & 2 (CCTT-1 & 2), Stroop test(color&word), Advanced test of attention, Wisconsin card sorting test, Korean - ADHD Rating Scale, to confirm Executive function. It can be judged by combining the results of each questionnaire test.
  This clinical trial, as an exploratory clinical trial, aims at seeing whether there is a statistical difference between before and after the treatment in observation items. If more than three are significant, the Executive function is considered significant.
Changes in Sleep disturbance | baseline, 2 weeks, 4 weeks
  Sleep disturbance is confirmed through the Korean version of the Children's Sleep Habits Questionnaire (K-CSHQ). This clinical trial, as an exploratory clinical trial, aims at seeing whether there is a statistical difference between before and after the treatment in observation items. This result is judged to be significant as the result value is lower.
Changes in Anxiety | baseline, 2 weeks, 4 weeks
  This is measured in two questionnaires, Korean Child Behavior Checklist (K-CBCL), The Korean version of State and Trait Anxiety Inventory for Children (K-STAIC), to confirm Anxiety. It can be judged by combining the results of each questionnaire test. The higher the score, the higher the Anxiety.
  This clinical trial, as an exploratory clinical trial, aims at seeing whether there is a statistical difference between before and after the treatment in observation items. If both items are significant, cognitive function is considered significant.
Changes in Sensory over - responsivity | baseline, 2 weeks, 4 weeks
  This is measured by Short Sensory Profile -2 (SSP-2) to confirm sensory over-responsivity. The higher the score, the higher the sensory over-responsivity. This clinical trial, as an exploratory clinical trial, aims at seeing whether there is a statistical difference between before and after the treatment in observation items. This result is judged to be significant as the result value is lower.
Changes in Clinical Global impression | baseline, 4 weeks
  This is determined through patient interviews. This clinical trial, as an exploratory clinical trial, aims at seeing whether there is a statistical difference between before and after the treatment in observation items. This result is judged to be significant as the result value is lower.

CONTACTS AND LOCATIONS:
Overall Officials: Hee Jeong Yoo, Ph. D., MD, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, South Korea

REFERENCES:
- [Derived] Han JH, Kim YR, Lee Y, Park Y, Kim D, Bong G, Yoo HJ. Double-blind, sham-controlled, pilot study of trigeminal nerve stimulation for autism spectrum disorder. Neurotherapeutics. 2026 Jan 29:e00838. doi: 10.1016/j.neurot.2026.e00838. Online ahead of print. PMID 41617599